CLINICAL TRIAL: NCT07131670
Title: A Prospective Observational Study on Symptom Burden in Lung Cancer Patients Undergoing Definitive Chemoradiotherapy: Insights From Electronic Patient-Reported Outcomes
Brief Title: Symptoms Burden in Lung Cancer Patients Undergoing Definitive Chemoradiotherapy: Insights From Electronic Patient-Reported Outcomes
Acronym: ePRO-LC-CRT
Status: Recruiting | Type: Observational
Sponsor: Qian Chu (Other)
Responsible Party: Sponsor-Investigator, Qian Chu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20240606
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Chemoradiotherapy; Patient-Reported Outcomes (PRO)
Keywords: Symptom Burden; Symptom Clusters; Electronic Patient-Reported Outcomes; MDASI-LC; Lung Cancer; EQ-5D
MeSH Terms: conditions — Lung Neoplasms; Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electronic Patient-Reported Outcome Monitoring — Participants complete the MDASI-LC and EQ-5D questionnaires electronically on a weekly basis during CRT and for 12 weeks after CRT. The data are used to evaluate symptom burden, symptom clusters, and symptom trajectories.

SUMMARY:
This prospective observational study aims to evaluate symptom burden and symptom clusters among lung cancer patients undergoing definitive concurrent chemoradiotherapy (CRT), based on electronic patient-reported outcomes (ePROs). Patients will complete the validated MDASI-LC and EQ-5D instruments weekly from baseline through the end of CRT and for 12 weeks post-treatment. The study will characterize the longitudinal trajectories of symptom severity and interference, identify distinct symptom clusters and their temporal patterns, and explore patient-level predictors of symptom burden. The findings may support the development of personalized symptom management strategies and improve quality of life during and after CRT.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed unresectable stage III NSCLC or limited-stage SCLC
* Age ≥ 18 years
* Receiving definitive chemoradiotherapy
* Able and willing to complete electronic questionnaires
* Provided written informed consent

Exclusion Criteria:

* Severe comorbidities (heart, liver, kidney)
* Psychiatric illness or cognitive impairment
* Prior chest or mediastinal radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients aged ≥18 years scheduled to receive definitive chemoradiotherapy at Tongji Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal trajectory of symptom burden over time based on M. D. Anderson Symptom Inventory-Lung Cancer | Baseline, weekly during CRT (weeks 1-6), and weekly for 12 weeks after CRT.
  M. D. Anderson Symptom Inventory-Lung Cancer:Scale range 0-10, with higher scores indicating worse symptom burden.

SECONDARY OUTCOMES:
Questionnaire response rate | From baseline to 12 weeks post-CRT
  The response rate of the M. D. Anderson Symptom Inventory-Lung Cancer( MDASI-LC) questionnaire will be assessed weekly during chemoradiotherapy (CRT) and up to 12 weeks post-CRT. This measure will reflect the percentage of patients who completed the MDASI-LC questionnaire each week, with higher response rates indicating better engagement and data quality.
Trajectory of symptom interference over time based on M. D. Anderson Symptom Inventory-Lung Cancer | From baseline to 12 weeks post-CRT
  M. D. Anderson Symptom Inventory-Lung Cancer: scale range 0-10, with higher scores indicating worse interference
Change of Quality of life over time | From baseline to 12 weeks post-CRT
  Quality of life will be assessed using the EuroQoL-5 Dimension Health Outcome Survey (EQ-5D) Questionnaire, a widely used instrument for measuring general health status. The EQ-5D includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The change in scores will be evaluated from baseline to 12 weeks after completion of chemoradiotherapy . Higher scores on the EQ-5D reflect better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

DOCUMENTS (1):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT07131670/Prot_000.pdf